CLINICAL TRIAL: NCT01711879
Title: Use of Intravitreal Aflibercept Injection for Neovascular Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-1526
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Neovascular Glaucoma
MeSH Terms: conditions — Glaucoma, Neovascular | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aflibercept with Laser (Active Comparator): A single injection of 2mg (0.05ml) intravitreal aflibercept injection at baseline followed by standard of care laser with observation for a total of 52 weeks
  Interventions: Drug: Aflibercept
- Aflibercept (Experimental): 2mg (0.05ml) intravitreal aflibercept injection at baseline followed by two additional injections at 4 weeks and 8 weeks, then every 8 weeks for a total of 52 weeks.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Details covered in arm description
  Other Names: Eylea

SUMMARY:
This 52 week study will assess the use of intravitreal aflibercept injections in patients with neovascular glaucoma (NVG) compared to standard of care panretinal photocoagulation.

The investigators hypothesize that the neovascularization of the iris and angle present in neovascular glaucoma will resolve more quickly in eye treated with intravitreal aflibercept injection alone and result in increased comfort and preservation of visual field as compared to current standard of care utilizing pan-retinal photocoagulation. The advantages to intravitreal aflibercept injection use could include resolution of NVI/NVA (neovascularization of the iris/neovascularization of the angle) leading to quicker pain relief and quicker lowering of IOP (intraocular pressure).

DETAILED DESCRIPTION:
The two arms of this study will compare current common practice (initial intravitreal anti-VEGF (vascular endothelial growth factor) to study treatment (VEGF) injection only) for 52 weeks.

This single center study will consist of 20 patients with NVG. Patients will be randomized to:

* Group A: A single injection of 2mg (0.05ml) intravitreal aflibercept injection at baseline followed by standard of care laser with observation for a total of 52 weeks.

or

* Group B: 2mg (0.05ml) intravitreal aflibercept injection at baseline followed by two additional injections at 4 weeks and 8 weeks, then every 8 weeks for a total of 52 weeks.

Clinical assessment will include pain assessment (Universal Pain Scale), best corrected visual acuity (ETDRS), ophthalmic examination, anterior segment assessment including number of clock-hours of NVI/NVA, gonioscopy, anterior segment photography, visual field test (Humphrey SITA- Standard 24-2), optic nerve OCT (Zeiss Cirrus Optic Disc Cube 200x200), macular OCT (Cube scan 512 x 128 and 5 Line Raster), fluorescein angiography (initial iris phase followed by standard retinal angiography), and concurrent medical/ocular medications. Qualitative assessment of neovascularization will be made by the investigator based on comparison to baseline angiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of neovascular glaucoma (Stage I-II)
* Individuals who are ages 21-90 years old; male or female of any race
* Presence of neovascularization of the iris and/or angle
* At least 90 degrees of "unzipped" anterior chamber angle as noted by gonioscopy. (a "zipped angle is the term used for a drainage angle that is slowly closing due to scar tissue from the neovascularization process)
* Visual acuity of light perception or better in the study eye
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent

Exclusion Criteria:

* Use of intravitreal anti-VEGF agents in the study eye in the past 3 months.
* Full PRP in the study eye
* Prior vitrectomy in the study eye
* Prior trabeculectomy or other filtration surgery in the study eye
* Active ocular or periocular infection in the study eye
* Ocular conditions (Cataract or vitreous hemorrhage) that might require surgery in next 12 months
* Allergy to fluorescein dye
* Any past use of systemic anti-VEGF medication
* Myocardial infarction within 6 months prior to study enrollment
* Stroke within 6 months prior to study enrollment
* Pregnant or breast-feeding women
* Sexually active men or women of childbearing potential who are unwilling to practice adequate contraception during the study

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malik Y Kahook, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Rocky Mountain Lions Eye Institute, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aflibercept With Laser | Aflibercept
Started | 3 | 4
Completed | 2 | 4
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept With Laser | Aflibercept | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.33 (5.69) | 61.5 (15.63) | 59.29 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Assess the safety profile of repeated intravitreal aflibercept injections in patients with NVG by evaluating the incidence of adverse events
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 3 | 4
Participants | 3 | 4

2. Primary Outcome: Severity of Adverse Events
Description: Assess the safety profile of repeated intravitreal aflibercept injections in patients with NVG by evaluating the severity of adverse events
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 3 | 4
Participants
  Abcess left thigh: Mild | 0 | 1
  Abcess left thigh: Moderate | 0 | 0
  Abcess left thigh: Severe | 0 | 0
  Abcess left thigh: None | 3 | 3
  Asthma: Mild | 0 | 1
  Asthma: Moderate | 0 | 0
  Asthma: Severe | 0 | 0
  Asthma: None | 3 | 3
  Pneumonia: Mild | 0 | 1
  Pneumonia: Moderate | 0 | 0
  Pneumonia: Severe | 0 | 0
  Pneumonia: None | 3 | 3
  Vitreous hemorrhage: Mild | 2 | 0
  Vitreous hemorrhage: Moderate | 0 | 0
  Vitreous hemorrhage: Severe | 0 | 0
  Vitreous hemorrhage: None | 1 | 4
  Worsening cataract non-study eye: Mild | 0 | 1
  Worsening cataract non-study eye: Moderate | 0 | 0
  Worsening cataract non-study eye: Severe | 0 | 0
  Worsening cataract non-study eye: None | 3 | 3
  Worsening Cataract Study eye: Mild | 1 | 1
  Worsening Cataract Study eye: Moderate | 1 | 0
  Worsening Cataract Study eye: Severe | 0 | 0
  Worsening Cataract Study eye: None | 1 | 3
  Diabetes Mellitus: Mild | 0 | 1
  Diabetes Mellitus: Moderate | 0 | 0
  Diabetes Mellitus: Severe | 0 | 0
  Diabetes Mellitus: None | 3 | 3
  Worsening NVG - non-study eye: Mild | 0 | 1
  Worsening NVG - non-study eye: Moderate | 0 | 0
  Worsening NVG - non-study eye: Severe | 0 | 0
  Worsening NVG - non-study eye: None | 3 | 3
  Recurrent BCC: Mild | 0 | 1
  Recurrent BCC: Moderate | 0 | 0
  Recurrent BCC: Severe | 0 | 0
  Recurrent BCC: None | 3 | 3
  progression of gall bladder cancer: Mild | 0 | 0
  progression of gall bladder cancer: Moderate | 0 | 0
  progression of gall bladder cancer: Severe | 1 | 0
  progression of gall bladder cancer: None | 2 | 4
  worsening of arthritis Right knee: Mild | 0 | 1
  worsening of arthritis Right knee: Moderate | 0 | 0
  worsening of arthritis Right knee: Severe | 0 | 0
  worsening of arthritis Right knee: None | 3 | 3
  matastatic cancer of liver: Mild | 0 | 0
  matastatic cancer of liver: Moderate | 0 | 0
  matastatic cancer of liver: Severe | 1 | 0
  matastatic cancer of liver: None | 2 | 4
  shortness of breath: Mild | 0 | 1
  shortness of breath: Moderate | 0 | 0
  shortness of breath: Severe | 0 | 0
  shortness of breath: None | 3 | 3

3. Secondary Outcome: Rate and Extent of Resolution of Neovascularization
Description: Compare between Groups A and B the Rate and extent of resolution of neovascularization in patients with NVG Stages 1 & 2.
Time Frame: 1 year
Population: No data was collected or analyzed for this Outcome Measure
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Intraocular Pressure (mmHg) at Baseline
Description: Intraocular pressure(mmHg) as measured by Goldmann applanation tonometry between groups A and B
Time Frame: Baseline
Population: One participant from group Aflibercept with Laser did not complete analysis due to death. Analysis is limited due to small sample size.
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 2 | 4
mmHg
  Study Eye Mean IOP(mmHg) at Baseline | 10 [08 to 12] | 23.5 [14 to 34]
  Fellow Eye Mean IOP(mmHg) at Baseline | 11 [08 to 14] | 22.75 [17 to 36]

5. Secondary Outcome: Intraocular Pressure (mmHg) at Week 52
Description: Mean intraocular pressure(mmHg) as measured by Goldmann applanation tonometry between groups A and B
Time Frame: Week 52
Population: as for outcome 4
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 2 | 4
mmHg
  Study Eye Mean IOP(mmHg) at W52 | 10 [08 to 12] | 15.25 [13 to 19]
  Fellow Eye Mean IOP(mmHg) at W52 | 10 [08 to 12] | 14 [06 to 20]

6. Secondary Outcome: Number of Patients Losing > 5 Letters on Visual Acuity in Each Group A and Group B
Description: Comparison between patients, groups A and B, that lost > 5 letters on visual acuity
Time Frame: Baseline to Week 52
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 3 | 3
participants | 0 | 0

7. Secondary Outcome: Number of Patients in Each, Group A and Group B, Gaining > 5 Letters on Visual Acuity
Description: Comparison of patients in each, group A and group B, that gained > 5 letters on visual acuity
Time Frame: Baseline to Week 52
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 3 | 3
participants | 2 | 0

8. Secondary Outcome: Visual Acuity at Baseline
Description: Comparison of visual acuity between groups A and B
Time Frame: Baseline
Population: as for outcome 4
Measure: Mean (Full Range); unit: Letters
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 2 | 4
Letters | 64 [64 to 64] | 37.5 [0 to 83]

9. Secondary Outcome: Visual Acuity at Week 52
Description: Comparison of visual acuity at Week 52 between groups A and B
Time Frame: Week 52
Population: as for outcome 4
Measure: Mean (Full Range); unit: Letters
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 2 | 4
Letters
  Study Eye Mean W52 Number of ETDRS Letters | 33.5 [0 to 67] | 62 [34 to 87]
  Fellow Eye Mean W52 Number of ETDRS Letters | 32 [0 to 64] | 46.75 [0 to 84]

10. Secondary Outcome: Comparison of the Visual Field Between Groups
Description: Comparison of the Visual field s measured by HVF 24-2 SITA Standards between groups A and B
Time Frame: 1 year
Population: No data was collected or analyzed for this Outcome Measure during the clinical trial.
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Measure of the Optical Coherence Tomography(OCT) Outcomes
Description: Evaluation of the Optical Coherence Tomography(OCT) outcomes (average retinal nerve fiber layer(RNFL) and central macular thickness), Compared between groups A and B.
Time Frame: Baseline to Week 52
Population: The database in OCT was corrupted and the data was lost
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Patients With Need for Surgical Intervention
Description: Comparison between groups A and B and the need for surgical intervention in both arms during the follow-up period
Time Frame: 1 year
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 3 | 3
participants | 0 | 0

13. Secondary Outcome: Number of Participants With Need for Additional IOP Lowering Medications
Description: Comparison between groups A and B for the need of additional IOP lowering medications
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 2 | 4
participants | 0 | 0

14. Secondary Outcome: Extent of Resolution of Neovascularization Between Groups
Description: Comparison of groups A and B and the extent of resolution of neovascularization in patients with NVG Stages 1 & 2
Time Frame: 1 year
Population: NVG Staging not recorded
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Evaluation of the Average Retinal Nerve Fiber Layer (RNFL)
Description: Comparison between groups A and B of the average retinal nerve fiber layer (RNFL) as measured by Optical Coherence Tomography (OCT)
Time Frame: 1 year
Population: The OCT database was corrupted and the data was lost
Arm/Group | Aflibercept With Laser | Aflibercept
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Aflibercept With Laser | Aflibercept
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept With Laser (N=3) | Aflibercept (N=4)
Death (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept With Laser (N=3) | Aflibercept (N=4)
Recurrent BCC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abcess left thigh (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vitreous hemmorrhage (Eye disorders) | 2 (2) | 0 (0)
Worsening cataract non-study eye (Eye disorders) | 0 (0) | 1 (1)
Worsening Cataract Study eye (Eye disorders) | 2 (2) | 1 (1)
Diabetes Mellitus (Endocrine disorders) | 0 (0) | 1 (1)
Worsening NVG - non-study eye (Eye disorders) | 0 (0) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
worsening arthritis right knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
progression of gall bladder cancer (Gastrointestinal disorders) | 1 (1) | 0 (0)
metastatic cancer affecting liver (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes